CLINICAL TRIAL: NCT03156244
Title: LCCC 1636: Using PROMIS as Part of Routine Clinical Care for Racially Diverse Prostate and Bladder Cancer Patients
Brief Title: Using PROMIS as Part of Routine Clinical Care for Racially Diverse Prostate and Bladder Cancer Patients
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1636
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer; Bladder Cancer
Keywords: PROMIS
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caucasian: This cohort will consist of 40 white patients who are receiving either radiation or surgery for treatment of their prostate or bladder cancer.
- African American: This cohort will consist of 40 African American patients who are receiving either radiation or surgery for treatment of their prostate or bladder cancer.

SUMMARY:
In this pilot study, a total of 80 patients with prostate or bladder cancer (40 black, 40 white) will complete 3 patient-reported outcome (PRO) surveys: baseline (pre-treatment), during treatment, and after treatment. The overall goal of this study is to assess whether collecting patient-reported data is feasible as part of clinical care of cancer patients, and whether these data are useful for clinicians and patients. Among these 80 patients, those who agree will also undergo a semi-structured interview to assess value of HRQOL assessment at the end of the study. Of specific interest is an evaluation of whether feasibility and perceived value differ between black and white participants.

DETAILED DESCRIPTION:
Cancer treatments, including surgery, radiotherapy and chemotherapy, are often linked to acute and late side effects. Historically, these effects were assessed by physicians and scored using standardized scales such as the Common Terminology Criteria for Adverse Events (CTCAE). Thorough and accurate assessment of symptoms facilitates timely and patient-centered symptom management.

Multiple studies have demonstrated that PROs more accurately capture patient symptoms than physician assessment. In a prospective trial, Falchook et al. investigated patient vs. physician report of symptoms in head and neck cancer patients undergoing radiotherapy (N=44). Patients and physicians separately completed weekly symptom assessments during treatment and once during follow-up. Patients tended to report more severe symptoms than physicians. For example, in week six, physicians rated 86% of patients' fatigue as non-existent or mild while 86% of patients rated their own fatigue as moderate to very severe. In a larger study conducted at Memorial Sloan-Kettering Cancer Center of 163 lung cancer patients undergoing chemotherapy, Basch et al. similarly examined patient vs. physician report of symptoms over one year. Compared to patients, physicians reported less severe and lower rates of fatigue, nausea, and pain and higher functional status.

Findings from these prior studies are consistent with evidence from a recent systematic review, which concluded that PRO data were essential for the evaluation of symptoms in cancer survivors. Many researchers have hypothesized the reasons behind this discrepancy in physician/patient ratings of symptoms, including poor communication, inadequate physician time spent per patient, and patients' underreporting of symptoms to physicians. Thus, incorporation of PRO data into routine clinical care can facilitate better detection and management of cancer and treatment-related effects.

Therefore, the goal of this pilot study is to move PRO data collection from a purely research exercise into using this as a tool to improve care for cancer patients. This pilot study will assess the feasibility of collecting PRO data as part of clinical care, and assess its "value" from the patient and physician perspectives. The investigators will recruit 80 patients with prostate or bladder cancers from the UNC Genitourinary Oncology clinics (including Urology and Radiation Oncology). PRO data that is most relevant to this patient population will be collected, including: gastrointestinal, urinary, sexual function, anxiety/depression, and sleep.

Further, given longstanding racial disparities in symptom experiences (e.g., symptom assessment, severity, frequency) among cancer patients and limited evidence of effective strategies for mitigating such inequities, this pilot study will also examine Black-White differences in terms of the feasibility and perceived value of sharing of patient-reported data to improve communication and decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Non-Hispanic Black and White patients with a known pathologic diagnosis of prostate or bladder cancer and intent to undergo treatment.
* Signed, IRB approved written informed consent.

Exclusion Criteria:

* Initiation of cancer-directed treatment
* Race/ethnicity other than Non-Hispanic Black or Non-Hispanic White
* Inability to read and speak English
* Inability to comply with study for any other reason than language
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A racially diverse cohort of 80 prostate and bladder cancer patients will be enrolled, including both male and female patients (n=40 Black; n=40 White) from the North Carolina Cancer Hospital's Multidisciplinary Urology and Radiation Oncology clinics
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of PRO assessments in a clinical setting | 90 days post treatment
  The feasibility of incorporating PRO assessments into the clinical setting for 80 Black and White patients undergoing treatment for bladder and prostate cancer. Feasibility is defined as at least 70% of study participants completing all three PRO assessments.

SECONDARY OUTCOMES:
Feasibility of enrollment | baseline
  The feasibility of enrolling bladder and prostate cancer patients into PRO assessment for clinical care. Feasibility of enrollment is defined as at least 37.56% of eligible patients who are approached about the study agree to enroll.
Preferred mode of questionnaire completion | baseline through 90 days post treatment
  The proportion of study participants who chose web vs. interactive voice response (IVR) as the preferred mode for PRO data collection. It is hypothesized 50% of patients will chose the web.
Feasibility by cohort | baseline through 90 days post treatment
  The rates of the feasibility of PRO assessment, the feasibility of enrollment, and preferred mode of PRO assessment in Black vs. White patients.
Perceived value | baseline through 90 days post treatment
  Patterns and Black vs. White differences in the perceived value of PRO assessments from the patient's perspective using semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Chen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Becky Green, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials